CLINICAL TRIAL: NCT03613025
Title: Performance of Non-targeted and/or Non-invasive Respiratory Samples for the Rapid Diagnosis of Pneumocystis Pneumonia Using the BDMAX TM Molecular Biology Platform (Becton Dickinson)
Brief Title: Non Invasive Diagnosis of Pneumocystis Pneumonia
Acronym: DANIPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC17.281; 2017-A02651-52 (Other: ID RCB)
Record Dates: First submitted 2018-07-09; First posted 2018-08-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pneumocystis
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case : confirmed PCP diagnosis (Other): Sampling of non-invasive and/or non-targeted respiratory tract specimens
  Interventions: Diagnostic Test: Sampling of non-invasive and/or non-targeted respiratory tract specimens
- Control : non confirmed PCP diagnosis (Other): Sampling of non-invasive and/or non-targeted respiratory tract specimens
  Interventions: Diagnostic Test: Sampling of non-invasive and/or non-targeted respiratory tract specimens

INTERVENTIONS:
Diagnostic Test: Sampling of non-invasive and/or non-targeted respiratory tract specimens — Sampling of oral fluids, sputa, bronchial aspiration in addition to BAL for the molecular diagnosis of PCP

SUMMARY:
Incidence and morbi-mortality of Pneumocystis pneumonia (PCP) are increasing. Early and fast diagnosis and treatment improve PCP prognosis. Biological diagnosis is based on the detection of Pneumocystis jirovecii, mainly by PCR, in broncho-alveolar lavage (BAL) obtained from bronchial fibroscopy. However this invasive exam is not always possible in emergency in suspected patient and others non invasive (sputa) and/or non-targeted (bronchial aspiration) are sent to the laboratory (25% of cases, data from the Grenoble University Hospital). Diagnosis performances of these non invasive/non-targeted samples are not clearly established.

In this study, the investigators aimed to establish the diagnosis value of non-invasive and/or non-targeted respiratory samples (oral fluids, sputa and bronchial aspiration) for the PCP diagnosis, compared to the gold-standard (Pneumocystis PCR on BAL, beta-D-glucans testing on serum and radio-clinical records).

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patient with (i) clinical and/or radiological suspicion of PCP, and (ii) bronchial fibroscopy with contributive BAL
* No immediate life-threatening conditions (estimated life expectancy >12h)
* No PCP treatment or PCP treatment < 48h
* Patient hospitalized in the Grenoble Alpes University Hospital with medical insurance
* Informed and written consent of the patient or its related

Exclusion Criteria:

* Pregnancy, breastfeeding
* Exclusion period of another clinical trial
* Deprivation of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 30 months
  Sensitivity of Pneumocystis PCR on non-invasive and/or non-targeted respiratory samples compared to the gold-standard
Specificity | 30 months
  Specificity of Pneumocystis PCR on non-invasive and/or non-targeted respiratory samples compared to the gold-standard
Area Under the Curve (AUC) | 30 months
  AUCs of Pneumocystis PCR on non-invasive and/or non-targeted respiratory samples compared to the gold-standard
Estimation of the positive predictive value | 30 months
  Estimation of the predictive values of Pneumocystis PCR on non-invasive and/or non-targeted respiratory samples compared to the gold-standard
Estimation of the negative predictive value | 30 months
  Estimation of the negative predictive values of Pneumocystis PCR on non-invasive and/or non-targeted respiratory samples compared to the gold-standard

SECONDARY OUTCOMES:
Time-saving (in hours) of PCP diagnosis on non-invasive and/or non-targeted respiratory samples compared to the PCP diagnosis on BAL, taking into account the time needed for bronchial fibroscopy | 30 months
Optimal cut-off values for interpretation of Pneumocystis fungal load on non-invasive and/or non-targeted respiratory samples | 30 months
Duration of anti-PCP treatment (days) | 30 months
  Impact of PCP diagnosis on non-invasive and/or non-targeted respiratory samples on the patient management
Estimation of the number of days of presumptive anti-PCP treatment that would have been avoided based on a PCP diagnosis on non-invasive and/or non-targeted respiratory samples | 30 months
  Impact of PCP diagnosis on non-invasive and/or non-targeted respiratory samples on the patient management
Estimation of the number of patients who would have received an earlier appropriate anti-PCP treatment based on a PCP diagnosis on non-invasive and/or non-targeted respiratory samples | 30 months
  Impact of PCP diagnosis on non-invasive and/or non-targeted respiratory samples on the patient management

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble Alpes University Hospital, Grenoble, France